CLINICAL TRIAL: NCT07398950
Title: Prospective Evaluation of Artificial Intelligence-enabled Screening for Transthyretin Amyloid Cardiomyopathy (ATTR-CM): TRACE-AI Prospective Study
Brief Title: Prospective Evaluation of Artificial Intelligence-enabled Screening for Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Acronym: TRACE-AI Yale
Status: Not yet recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Bridgebio Pharma, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000039677
Record Dates: First submitted 2025-07-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ATTR Amyloidosis With Cardiomyopathy; Heart Failure
Keywords: Transthyretin Amyloid Cardiomyopathy (ATTR-CM); Artificial Intelligence Screening; AI-ECG; AI-Echo; Electrocardiogram; Technetium-99m Pyrophosphate (Tc99m-PYP) Scintigraphy; Machine Learning in Cardiology; Validation of AI Diagnostic Tools; Cardiomyopathy Screening; Early Detection of Cardiac Amyloidosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ATTR-CM AI-ECG and AI-Echo Model — AI-based sequential screening approach for ATTR-CM

SUMMARY:
The TRACE-AI Diagnostic Study will evaluate the performance of artificial intelligence (AI) models applied to electrocardiograms (AI-ECG) and echocardiograms (AI-Echo) to identify transthyretin amyloid cardiomyopathy (ATTR-CM) in adults with heart failure. Model performance will be validated through comparison with technetium-99m pyrophosphate (PYP) imaging results.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with at least one of each component cardiovascular diagnosis testing (ECG and Echo) in the YNHHS.
* Patients with a diagnosis of HFpEF or HFmrEF
* Participant from Phase I TRACE-AI Study with AI-ECG and AI-Echo screen in the preceding 36 months

Exclusion Criteria:

* Patients who have opted out of research studies
* Patients with cardiac amyloid diagnostic test in the past 36 months
* Patients with hypertrophic cardiomyopathy or end-stage renal disease
* Pregnant women
* Patients unable or unwilling to provide informed consent
* Non-English speakers and cognitively impaired individuals who are unable to comprehend the consent and the on-screen instructions on the application, which are in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants from the YNHHS who were identified in Phase I of the TRACE-AI study. Eligible individuals must have a confirmed diagnosis of HFpEF or HFmrEF, 75 with a positive AI-based screening result from both AI-ECG and AI-Echo and 75 with a negative AI-based screen, and no prior diagnostic work-up for cardiac amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Performance of the sequential screening approach | From enrollment through completion of PYP scan at baseline study visit
  Measured by the positive predictive value (PPV) of the test for ATTR-CM, based on confirmatory imaging and clinical testing

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Khera, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No